CLINICAL TRIAL: NCT03411811
Title: Dextrose Prolotherapy in Chronic Ulnar Wrist Pain Resistant to Usual Care: Comparison to a Naive-to-treatment Cohort Who Receive Usual Care
Brief Title: Ulnar Wrist Pain Treatment With Dextrose Prolotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Abierta Interamericana (Other)
Collaborators: Gonzaolo Yaumauchi, M.D. (Unknown)
Responsible Party: Principal Investigator, Ezequiel Mailand and Miguel Slullitel, Ezequiel Mailand, M.D., Principal Investigator., Universidad Abierta Interamericana
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UniversidadAI
Record Dates: First submitted 2018-01-03; First posted 2018-01-26 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Ulnar Wrist Pain
Keywords: tendinopathy; wrist; chronic pain; sprain
MeSH Terms: conditions — Tendinopathy; Chronic Pain; Sprains and Strains | interventions — Glucose

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel. After that the study becomes one arm as both groups are offered dextrose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator)
  Interventions: Other: Usual Care
- Dextrose (Experimental)
  Interventions: Procedure: Dextrose

INTERVENTIONS:
Other: Usual Care — Therapeutic ultrasound, myofascial release of extensor and flexor muscles of forearm and stabilization exercises for the wrist.
  Arms: Usual Care
Procedure: Dextrose — Injection of 1 ml of 12.5% dextrose in 1% lidocaine at 0, 3 and 6 weeks in 5 locations: Origin of ulnar collateral ligament, insertion of ulnar collateral ligament on the triquetrum, insertion of the extensor carpi ulnaris on the base of the 5th metacarpal, triquetral hamate ligament and ulnotriquetral joint space.
  Arms: Dextrose

SUMMARY:
Participants who have failed therapy for chronic wrist pain on the little finger side of the wrist will recieve dextrose prolotherapy. Their results will be compared to a cohort of consecutive participants who have not failed therapy, and receive 4 weeks of usual care.

ELIGIBILITY:
Inclusion criteria

* Pain on the ulnar side of the wrist.
* PRWE greater than 40

Exclusion criteria

* Radioulnar instability more than moderate as determined by a positive ulna fovea sign or ulna grinding test
* Surgery in the wrist area
* Infection in the wrist area
* Other wrist pathology on examination
* Other pain area that is constant, interferes with sleep, or is as bad, or worse, than shoulder pain.
* Diabetes or other peripheral neuropathy
* Radiculopathy
* Unstable psychiatric function.
* Current opioid use.
* Vulnerable patients
* Pregnancy

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline PRWE (Patient Rated Wrist Evaluation) at 9 weeks | 9 weeks
  The PRWE is a 15-item questionnaire designed to measure wrist pain and disability in activities of daily living.
Change from baseline PRWE between 0 weeks and 1 year | 1 year
Percentage of participants exceeding a PRWE change of plus 14 between baseline and 9 weeks | 9 weeks
Percentage of participants exceeding a PRWE change of plus 14 between baseline and 1 year | 1 year

SECONDARY OUTCOMES:
Satisfaction score at 9 weeks | 9 weeks
  On a scale from 1-5 please rate satisfaction with your results. 1 means 'no satisfaction' and 5 means 'complete satisfaction'.
Satisfaction score at 1 year | 1 year
  On a scale from 1-5 please rate satisfaction with your results. 1 means 'no satisfaction' and 5 means 'complete satisfaction'

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Slullitel, M.D., Principal Investigator — Universidad Abierta Interamericana
Locations (1):
- Scanner Centro de Diagnostico, Rosario, Santa Fe Province, Argentina

IPD SHARING:
Plan to Share IPD: Undecided
Anticipate sharing data by request

REFERENCES:
- [Background] Tay SC, Tomita K, Berger RA. The "ulnar fovea sign" for defining ulnar wrist pain: an analysis of sensitivity and specificity. J Hand Surg Am. 2007 Apr;32(4):438-44. doi: 10.1016/j.jhsa.2007.01.022. PMID 17398352
- [Background] Spies CK, Muller LP, Oppermann J, Hahn P, Unglaub F. [Instability of the distal radioulnar joint - an overview of clinical and radiological procedures regarding their efficacies]. Handchir Mikrochir Plast Chir. 2014 Jun;46(3):137-50. doi: 10.1055/s-0033-1363662. Epub 2014 Feb 18. German. PMID 24549807
- [Background] Reeves KD, Sit RW, Rabago DP. Dextrose Prolotherapy: A Narrative Review of Basic Science, Clinical Research, and Best Treatment Recommendations. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):783-823. doi: 10.1016/j.pmr.2016.06.001. PMID 27788902